CLINICAL TRIAL: NCT06412016
Title: ProMeSA: Urban Gardening and Peer Nutritional Counseling to Improve HIV Care Outcomes Among People With Food Insecurity in the Dominican Republic
Brief Title: Urban Gardening and Peer Nutritional Counseling for People With HIV and Food Insecurity
Acronym: ProMeSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of California, San Francisco (Other); Universidad Autonoma de Santo Domingo (Unknown); CONAVIHSIDA, Republica Dominicana (Unknown); Ministerio de Agricultura, Republica Dominicana (Unknown); Ministerio de Salud Publica y Asistencia Social, Republica Dominicana (Other Government); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01MH131447 (NIH)
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: HIV; Food Insecurity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analytic database will not have any indication of intervention or control group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Nutritional Counseling + Urban Gardening (Experimental): Participants in the intervention clinics will receive: 1) nutritional counseling from peer counselors in their clinic (4 sessions administered); 2) training from the Ministry of Agriculture on how to plant and maintain a garden in their home (2 group training workshops and monthly individual follow-up); 3) low-cost tanks for water storage to participants whose communities only have water on certain days; 4) access to community gardens; and 5) two cooking and nutrition workshops.
  Interventions: Behavioral: Peer Nutritional Counseling + Urban Gardening
- Usual Care Control (No Intervention): Participants in the control clinics will receive their usual care from the clinic. After 18-month follow-up, they will be offered the opportunity to receive the intervention.

INTERVENTIONS:
Behavioral: Peer Nutritional Counseling + Urban Gardening — Peer nutritional counseling and urban gardens
  Arms: Peer Nutritional Counseling + Urban Gardening

SUMMARY:
The investigators are conducting a fully powered cluster randomized controlled trial (RCT) of a culturally appropriate, multicomponent intervention combining peer nutritional counseling with urban gardening among people with human immunodeficiency virus (HIV) in the Dominican Republic (DR) to assess efficacy, analyze mediators of effects, and evaluate detailed process data to inform scale-up. The study will examine the impact of the intervention on participants' HIV clinical outcomes (HIV viral load, antiretroviral therapy adherence, and HIV care retention) as well as intermediate outcomes such as food security and HIV-related stigma.

DETAILED DESCRIPTION:
HIV and food insecurity pose severe and interrelated problems in Latin America and the Caribbean, including in the Dominican Republic (DR), where HIV ranks as one of the top 5 causes of death and our prior studies have found that nearly 70% of people with HIV (PWH) have moderate or severe food insecurity. Despite the established, detrimental role of food insecurity on poor HIV treatment outcomes, evidence on sustainable interventions that address the cycle of food insecurity and poor HIV health is scarce. To address this gap, the investigators developed and piloted Proyecto para Mejorar la Seguridad Alimentaria (ProMeSA or Project to Improve Food Security in English), an integrated urban gardens and peer nutritional counseling intervention, and found it feasible, acceptable, and with preliminary efficacy at 6 and 12 months of improving food security and HIV virologic suppression. The purpose of this 5-year study is to conduct a fully powered cluster randomized controlled trial (RCT) of ProMeSA to assess intervention efficacy evaluated over a longer period (18 months) as well as mediators and barriers and facilitators to intervention uptake, implementation, and sustainability. The specific aims are: (1) Determine the efficacy of an integrated urban gardens and peer nutritional counseling intervention on the primary outcome of HIV viral suppression [undetectable HIV viral load (VL)] and secondary outcomes of antiretroviral therapy (ART) adherence and HIV care retention care among people with food insecurity across diverse regions in the DR; (2) Examine the intervention effects on intermediate outcomes posited to mediate the impact of ProMeSA on ART adherence, care retention, and viral suppression; (3) Evaluate process-related factors associated with intervention uptake and implementation (facilitators, barriers, fidelity, and replication costs) to inform future scale-up. The trial will include 20 HIV clinics randomized to intervention or usual care control (n=25 per clinic; *500 total study participants). VL and other key outcomes will be assessed at baseline, and 6-, 12- and 18-months. Following the investigators' intervention causal framework and pilot findings, they hypothesize that ProMeSA will improve food security and diet quality and reduce stigma and competing needs, which in turn will improve HIV clinical outcomes. The predominant causal paths identified will inform tailoring ProMeSA to enhance impact in future dissemination and implementation. In addition, the investigators will collect extensive quantitative and qualitative data on intervention implementation and participant experiences with the intervention across diverse settings and participants to inform scale-up. The study involves a partnership among researchers from the University of Massachusetts Amherst, University of California, San Francisco, RAND, and the Universidad Autonóma de Santo Domingo as well as the Dominican Ministries of Agriculture and Public Health, the Dominican National HIV/AIDS Council, and the United Nations World Food Program. To the investigators' knowledge, this will be the first full-scale trial to integrate nutritional counseling with food-generating activities among PWH with food insecurity, in support of national and international goals to achieve viral suppression and reduce the disease- and economic burden of HIV. [*Update: Because of recruitment challenges at some clinics due to USAID funding cuts and lower detectable viral load, we received NIH approval to reduce sample size to n=433 while retaining similar power]

ELIGIBILITY:
Inclusion Criteria:

1. registered at one of the 20 HIV clinics in the study;
2. age 18 or older;
3. having initiated ART at least 6 months ago;
4. detectable viral load in the previous 12 months based on medical records and/or evidence of adherence problems (missed clinic visits, delays in picking up antiretrovirals);
5. moderate or severe household food insecurity
6. physically able to plant and maintain an urban garden; stable housing and space for a garden (subjectively assessed by participants after hearing a description of what is involved)
7. planned residency in the local area for the duration of the study

Exclusion Criteria:

Does not meet above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HIV viral load | Change in viral load between baseline and months 6, 12, and 18
  Change in viral load

SECONDARY OUTCOMES:
Antiretroviral therapy adherence | 6, 12 and 18 months
  Self-reported adherence and objective adherence verified through pharmacy refills
HIV care retention | 6, 12, and 18 months
  Self-reported missed clinic visits verified through clinic records

OTHER OUTCOMES:
Food Insecurity | 6, 12 and 18 months
  Self-reported food security using the Latin American and Caribbean Food Security Scale to assess household food security over the past 90 days. Scores range from 0 to 15 for households with children (0-8 for households without children) with higher scores meaning worse outcome and are used to classify households into 4 categories: "food secure," "mild food insecurity, "moderate food insecurity" and "severe food insecurity."
Internalized HIV Stigma | 6, 12 and 18 months
  Self-reported internalized stigma will be assessed using an 8-item scale validated previously in the DR. Answers use a 4-point Likert scale (strongly disagree to strongly agree) assessing agreement with statements measuring negative self-perceptions related to HIV; higher scores indicated worse internalized stigma, range 0-32.
Experienced HIV Stigma (Discrimination) | 6, 12 and 18 months
  Self-reported experienced stigma will be assessed using 11 items on reported loss of job, denial of health and other social services, and being verbally harassed or physically abused as a result of living with HIV (with responses of "yes/no"). This scale been validated in the DR previously and examined both as continuous (range 0-11, with higher scores meaning worse outcome) and dichotomously (any experienced stigma vs. none).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn P Derose, PhD, MPH, Principal Investigator — University of Massachusetts, Amherst
Locations (20):
- Dominican Republic (20):
  - Hospital Taiwan 19 de marzo, Azua
  - Hospital Nuestra Señora de la Altagracia, Higüey
  - CPN Las Cinco Casas, Monte Plata
  - Hospital Nuestra Señora de Regla, Peravia
  - Hospital Ricardo Limardo, Puerto Plata
  - SAI Veron, Punta Cana
  - Hospital Leopoldo Pou, Samaná
  - Hospital Juan Pablo Pina, San Cristóbal
  - Hospital San Vicente de Paul, San Francisco de Macorís
  - Hospital Dr. Alejandro Cabral, San Juan de la Maguana
  - Centro de Salud Integral Bella Vista, Santiago de los Caballeros
  - Centro Especializado de Atención de Salud Juan XXIII, Santiago de los Caballeros
  - Hospital José María Cabral y Báez, Santiago de los Caballeros
  - Instituto Dominicano de Estudios Virológicos IDEV, Santo Domingo
  - Centro Sanitario de Santo Domingo, Santo Domingo
  - Hospital Dr Luis Eduardo Aybar, Santo Domingo
  - SAI Activo 20-30, Santo Domingo
  - Centro de Orientación e Investigación Integral COIN, Santo Domingo
  - AID for AIDS-Tu Salud, Santo Domingo Este
  - Hospital Dr. Vinicio Calventi, Santo Domingo Oeste

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported, biometric, chart abstraction, pharmacy refill, and clinical outcome variables. Following publication of the main paper(s) for this study and the grant end-date, the investigators will make the data publicly available in the form of an electronic database for researchers who successfully complete a registration process. Data will be de-identified and will not contain any direct identifiers or indirect identifiers. The investigators will provide documentation in the form of a codebook in which each variable name and response options are defined. As part of the registration process, users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.
Supporting Information: SAP
Time Frame: Data will become available after publication of study results, approximately 2032 for five years
Access Criteria: Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the public use dataset.